CLINICAL TRIAL: NCT01893073
Title: Effectiveness of a a Mindful Walking Program in Patients With Chronic Low Back Pain - a Randomized Controlled Trial
Brief Title: Mindful Walking in Low Back Pain
Acronym: MW-LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Benno Brinkhaus, Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MW-LBP
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Low Back Pain

ARMS (2):
- Mindful walking (Active Comparator): A weekly 60 minutes walking group exercise program consisting of a combination of walking and mindfulness over 8 weeks.
  Interventions: Behavioral: Mindful walking program
- Waiting group (No Intervention)

INTERVENTIONS:
Behavioral: Mindful walking program
  Arms: Mindful walking

SUMMARY:
The purpose of this study is to determine whether a mindful walking program is effective in the treatment of patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* male and female, 18-65 years
* chronic low back pain (disease duration > 3 months)
* pain intensity on visual analogue scale at inclusion > 40 mm (0-100 mm scale)
* only pharmacological treatment with NSAID or no treatment in the last 4 weeks
* undersigned informed consent form

Exclusion Criteria:

* active walking or jogging in the last 6 weeks (< 60 minutes/week)
* regular meditation, relaxation exercise, mindfulness exercise in last 6 weeks (> 30 minutes per week)
* use of complementary medicine therapies as acupuncture, homeopathy, herbal medicine in last 6 weeks or planned in the next 12 weeks
* use of other nonpharmacological therapies as physical therapy, manual therapy or osteopathy in the last 4 weeks
* participation in another trials within the last 3 months
* pathological neurological symptoms such as muscular paralysis or paraesthesia due to spinal disc herniation or other causes
* risk of falls and inability to walk
* angina pectoris in the last 3 months
* chronic respiratory disease with respiratory insufficiency
* intake of central nervous system-acting analgesics in the last 6 weeks
* Known renal and / or hepatic diseases
* Severe organic, psychological or psychiatric disorders that are not permitting a study participation
* applying for early retirement due to low back pain
* no undersigned informed consent form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity on visual analogue scale | 8 weeks

SECONDARY OUTCOMES:
Back function - FFbH-R-Questionnaire | 8 weeks, 12 weeks
Pain intensity on visual analogue scale | 12 weeks
Cohens perceived stress scale | 8 weeks, 12 weeks
Quality of Life - SF 36 | 8 weeks, 12 weeks
Intake of paracetamol | 8 weeks
Adverse events | 8 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Social Medicine, Epidemiology and Health Economics, Charité Universitätsmedizin Berlin, Germany, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Rotter G, Ortiz M, Binting S, Tomzik J, Reese F, Roll S, Brinkhaus B, Teut M. Mindful Walking in Patients with Chronic Low Back Pain: A Randomized Controlled Trial. J Integr Complement Med. 2022 Jun;28(6):474-483. doi: 10.1089/jicm.2021.0361. Epub 2022 Mar 30. PMID 35363058